CLINICAL TRIAL: NCT00681993
Title: "A Feasibility Trial of Partial Breast Irradiation With Various Concurrent Chemotherapy Regimens (PBIC)"
Brief Title: Trial of Partial Breast Irradiation With Various Concurrent Chemotherapy Regimens
Acronym: PBIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0805; IRB00063221 (Other: JHM IRB)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: cosmetic; effect; breast; irradiation; concurrent; chemotherapy; potential acute; late skin; subcutaneous toxicities
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; carboxypeptidase M; Carboplatin; Trastuzumab; Docetaxel; Receptor Protein-Tyrosine Kinases; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Standard ddAC chemotherapy with concurrent radiation therapy (Active Comparator): Standard dose-dense Adriamycin and Cyclophosphamide (ddAC) chemotherapy and concurrent radiation therapy (RT)
  Interventions: Other: Standard Dose Dense Doxorubucin and Cyclophosphamide
- Standard AC chemotherapy with concurrent RT (Active Comparator): Standard Adriamycin and Cyclophosphamide (AC) chemotherapy and concurrent radiation therapy
  Interventions: Other: Standard Doxorubucin and Cyclophosphamide
- Standard TCarbo H chemotherapy with concurrent RT (Active Comparator): Standard Taxotere, Carboplatin and Herceptin (TCarbo H) chemotherapy and concurrent radiation therapy
  Interventions: Other: Standard Docetaxel, Carboplatin, and Herceptin
- Standard TAC chemotherapy with concurrent RT (Active Comparator): Standard Taxotere, Adriamycin and Cyclophosphamide (TAC) chemotherapy with concurrent radiation therapy
  Interventions: Other: Standard Docetaxel, Doxorubucin and Cyclophosphamide
- Standard TC chemotherapy with concurrent RT (Active Comparator): Standard Taxotere and Cyclophosphamide (TC) chemotherapy with concurrent radiation therapy
  Interventions: Other: Standard Docetaxel and Cyclophosphamide

INTERVENTIONS:
Other: Standard Dose Dense Doxorubucin and Cyclophosphamide — 4 cycles of Standard Dose-Dense Doxorubucin and Cyclophosphamide and concurrent radiation therapy at a dose of 270 cGy per fraction for 15 fractions to a total dose of 40.5 Gy. Treatments will be given Monday through Friday for three weeks. Radiation therapy may start 7 days before, but no later than 7 days after, day 1 of cycle 1 of chemotherapy (C1D1).
  Other Names: Doxorubucin (Adriamycin, Rubex, Adriamycin RDF, Adriamycin PFS,; hydroxydaunorubicin, hydroxydaunomycin); Cyclophosphamide (Cytoxan, Neosar, CTX, CPM)
  Arms: Standard ddAC chemotherapy with concurrent radiation therapy
Other: Standard Doxorubucin and Cyclophosphamide — 4 cycles of Standard Dose Doxorubucin and Cyclophosphamide and concurrent radiation therapy at a dose of 270 cGy per fraction for 15 fractions to a total dose of 40.5 Gy. Treatments will be given Monday through Friday for three weeks. Radiation therapy may start 7 days before, but no later than 7 days after, day 1 of cycle 1 of chemotherapy (C1D1).
  Other Names: Doxorubucin (Adriamycin, Rubex, Adriamycin RDF, Adriamycin PFS,; hydroxydaunorubicin, hydroxydaunomycin); Cyclophosphamide (Cytoxan, Neosar, CTX, CPM)
  Arms: Standard AC chemotherapy with concurrent RT
Other: Standard Docetaxel, Carboplatin, and Herceptin — 6 cycles of Standard Docetaxel, Carboplatin and Herceptin chemotherapy with concurrent radiation therapy at a dose of 270 cGy per fraction for 15 fractions to a total dose of 40.5 Gy. Treatments will be given Monday through Friday for three weeks. Radiation therapy may start 7 days before, but no later than 7 days after, day 1 of cycle 1 of chemotherapy (C1D1).
  Other Names: Docetaxel (Taxotere); Carboplatin (CBDCA, Paraplatin, JM-8); Herceptin (Trastuzumab, RhuMAb HER2, HER2/neu, anti-HER2 humanized; monoclonal antibody)
  Arms: Standard TCarbo H chemotherapy with concurrent RT
Other: Standard Docetaxel, Doxorubucin and Cyclophosphamide — 3 cycles of Standard Docetaxel, Doxorubucin and Cyclophosphamide chemotherapy with concurrent radiation therapy at a dose of 270 cGy per fraction for 15 fractions to a total dose of 40.5 Gy. Treatments will be given Monday through Friday for three weeks. Radiation therapy may start 7 days before, but no later than 7 days after, day 1 of cycle 1 of chemotherapy (C1D1).
  Other Names: Docetaxel (Taxotere); Cyclophosphamide (Cytoxan, Neosar, CTX, CPM)
  Arms: Standard TAC chemotherapy with concurrent RT
Other: Standard Docetaxel and Cyclophosphamide — 4 cycles of Standard Docetaxel and Cyclophosphamide chemotherapy with concurrent radiation therapy at a dose of 270 cGy per fraction for 15 fractions to a total dose of 40.5 Gy. Treatments will be given Monday through Friday for three weeks. Radiation therapy may start 7 days before, but no later than 7 days after, day 1 of cycle 1 of chemotherapy (C1D1).
  Other Names: Docetaxel (Taxotere); Cyclophosphamide (Cytoxan, Neosar, CTX, CPM)
  Arms: Standard TC chemotherapy with concurrent RT

SUMMARY:
Breast conserving therapy, (BCT), which consists of wide local excision of the tumor followed by 6 weeks of whole breast irradiation, (WBI), is integral to the management of breast cancer. Evidence now suggests that WBI may not be necessary and treatment to the involved area only, partial breast irradiation, (PBI), may suffice. PBI can be achieved by interstitial or intracavitary brachytherapy, intra-op, or post op external beam radiation therapy. The feasibility, toxicity and efficacy of PBI are currently being studied in both the U.S. and Europe. Review of smaller studies suggests that PBI will prove to be comparable to WBI. Chemotherapy combined with radiation has been shown to increase local control in BCT when compared to radiation alone. However there is little data on how sequencing or timing of these therapies with respect to one another affect outcome. As a result there is no consensus about the optimal combination. There are real and potential benefits to concurrent chemo-radiation therapy. Concurrent therapy 1) allows both treatments to start closer to surgery, theoretically maximizing the benefits of each modality; 2) shortens the overall treatment program; and 3) may also improve local control via chemo-sensitization of residual cancer cells. However, concurrent chemotherapy and WBI have been associated with prohibitive skin toxicity. Since less breast tissue is treated with PBI, this skin toxicity may no longer be prohibitive. We have shown in J0381 that PBI and concurrent dose dense AC is safe. As a follow-up, we propose a phase I/II trial addressing the toxicity and efficacy associated with PBI delivered concurrently with various chemotherapy regimens.

DETAILED DESCRIPTION:
1. Partial Breast Irradiation with concurrent chemotherapy (various regimens. Subjects will receive Segmental Mastectomy (Lumpectomy)
2. Medical Oncology Evaluation
3. Consent/Registration Pre-RT evaluation
4. Simulation/Treatment Planning
5. Chemo-Radiation Therapy:

   ddAC, Std AC, TAC, TC, TCH or TH Concurrent with PBI - (270 cGy per fraction for 15 fractions). RT may start up to 7days prior to C1D1, but no later than 7 days after C1D1 (+/- 7 days of C1D1 radiation may start)
6. Further chemotherapy, hormonal therapy or biologic therapy at the medical oncologist's discretion
7. F/U Schedule

ELIGIBILITY:
Eligibility Criteria:

Each of the criteria in the following section must be met in order for a patient to be considered eligible for registration.

* Patient must be older than 18 years of age
* Patients must have histologically confirmed (by routine H&E staining) adenocarcinoma of the breast, with the primary tumor < 4 cm and 0 - 3 positive axillary lymph nodes (pathologic T1-2, pathologic N0 -N1, M0). Patients with squamous carcinomas or sarcomas of the breast cancer are NOT eligible.
* Patient must have a history and physical within six weeks prior to the start of any protocol therapy.
* Patient must have had a bilateral mammogram prior to surgery.
* Patients must have undergone a segmental mastectomy (SM) with a level I and ll axillary dissection or sentinel lymph node biopsy. Surgical margins at time of SM must be negative (> or = 2 mm) for both invasive carcinoma and for non-invasive ductal carcinoma. Patients who have post-operative margins which are negative but less than 2mm will be considered eligible if the surgeon states that the margin in question could not be improved.
* Patient must have a Medical Oncology consult and be recommended to receive one of the following regimens: Cyclophosphamide and Doxorubicin (AC); Taxotere, Doxorubicin and Cyclophosphamide (TAC); Taxotere and Cyclophosphamide (TC) or Taxotere, Carboplatin and Trastuzumab (TCH) prior to registration. The use of additional chemotherapy, hormonal therapy or Trastuzumab after the initial regimen is at the discretion of the medical oncologist.
* Patients must be registered such that radiation therapy begins no sooner than 7 days prior to, but no later than 7 days after, day 1 of cycle 1 (C1D1). Patient must start chemotherapy and radiation less than 14 weeks from the last breast surgical procedure.
* Patients must NOT have received any neo adjuvant chemo or hormonal therapy for the current cancer.
* Patients must have a performance status 0 or 1 by ECOG criteria
* Patients must not have received prior radiation therapy to the involved breast at any time for any reason.
* Any patient with active local-regional disease prior to registration is not eligible.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for 5 years.
* Patients must not be pregnant due to the potential for fetal harm as a result of this treatment regimen. Women of child-bearing potential must use effective non hormonal contraception while undergoing radiation therapy. Women of child-bearing potential must also have a negative pregnancy test within six weeks prior to start of protocol therapy.
* Patients must not have a serious medical or psychiatric illness which prevents informed consent or compliance with treatment.
* All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2016-03-04 (Actual)

PRIMARY OUTCOMES:
Acute skin toxicities of partial breast irradiation concurrent with chemotherapy (PBIC) | up to 5 years post-intervention
  Acute Skin toxicity will be scored on a scale ranging from 0-4, where a higher score reflects more severe toxicity:
  0= no change; 1= follicular, fain or dull erythema/epilation/dry/desquamation/decreased swelling; 2= tender or bright erythemal patchy moist desquamation/moderate edema; 3= confluent moist desquamation other than skin folds, pitting edema; 4= ulceration, hemorrhage, necrosis.
Late skin toxicities of PBIC | up to 5 years post-intervention
  Late Skin toxicity will be scored on a scale ranging from 0-4, where a higher score reflects more severe toxicity:
  0= none; 1= slight atrophy, pigmentation change, some hair loss; 2= patchy atrophy, moderate telangiectasias, total hair loss; 3= marked atrophy, gross telangiectasias; 4= ulceration
Subcutaneous tissue toxicities of PBIC | up to 5 years post-intervention
  Subcutaneous tissue toxicity will be scored on a scale ranging from 0-4, where a higher score reflects more severe toxicity:
  0= none; 1= slight induration (fibrosis) and loss of subcutaneous fat; 2= moderate fibrosis but asymptomatic; slight field contracture; <10% linear reduction; 3= severe induration and loss subcutaneous tissue; field contracture >10% linear reduction; 4= necrosis

SECONDARY OUTCOMES:
Cosmetic effect of PBIC | up to 5 years post-intervention
  Number of participants with Poor, Fair, Good, or Excellent cosmetic effect after PBIC. Cosmetic effect will be graded by the investigator and participant as specified by the grading criteria in the Study Protocol (grading criteria description too large for this field).
Local control rate of patients treated with PBIC. | up to 5 years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zellars, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Amit Shah, M.D., Principal Investigator — York Cancer Center
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States